CLINICAL TRIAL: NCT01913197
Title: Phase I/II Evaluation Magnetic Resonance Imaging (MRI)-Guided Differential-Dose Prostate Brachytherapy
Brief Title: Using Magnetic Resonance Imaging (MRI) to Guide Differential-Dose Prostate Brachytherapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-070
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Brachytherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pre-implant MRI images and planning (Experimental)
  Interventions: Other: An MRI-based technique to identify prostate cancer

INTERVENTIONS:
Other: An MRI-based technique to identify prostate cancer

SUMMARY:
In standard prostate brachytherapy treatment, the seeds are placed throughout the prostate to treat the entire gland. This is done because, in the past, it was impossible to know where the cancer was located within the prostate. Multiparametric magnetic resonance imaging (MRI) can identify tumor(s) with a high degree of accuracy. This trial will assess whether using MRI to guide prostate brachytherapy can result in less chronic toxicity by allowing lower doses to be delivered to the regions of the prostate without tumor while simultaneously allowing higher doses to the tumor. Subjects enrolled in this study will then be followed over two years and evaluated for toxicity. In addition, after two years they will undergo an MRI and a biopsy to assess the cancer control rate of the treatment.

DETAILED DESCRIPTION:
Prostate brachytherapy is a popular treatment for clinically localized prostate cancer. In properly selected patients, it is highly effective with biochemical (PSA) disease free survival rates of 85-95% at 5-10 years. However, the technique is currently limited by the inability to localize the cancer within the prostate. The multifocal nature of prostate cancer is well established. Because of the inability to know where within the prostate the cancer is located, radiation must be delivered throughout the gland. Although this blind approach leads to good results, it is clear that there are regions of the prostate and surrounding tissue that are overexposed to radiation while others are underexposed relative to their true need based on their tumor burden and their proximity to the tumor areas. Multiple studies have shown significant correlation between MRI abnormalities and radical prostatectomy specimens for determining size and location of cancer foci. MRI images have already begun to be incorporated into diagnostic and therapeutic procedures for prostate cancer on an experimental basis by other investigators. The images have been fused with real time TRUS to successfully perform targeted biopsies. In this study, we propose to use MRI images in the pre-treatment planning process to identify the tumors within the prostate prior to the brachytherapy and use these images to direct the dosimetry planning. The primary goal of this study is to decrease the chronic toxicities as assessed by the Common Toxicity Criteria Version 4.0 by decreasing the integral dose to the regions of the prostate which do not have tumor. A secondary goal is to increase the dose to the tumor(s) and demonstrate this ability while maintaining the urethral and other normal tissue doses. We also wish to perform dosimetric comparisons of the normal tissues and the tumor(s) when this technique is used compared to what would have been done if the patient had received a traditional implant. Finally, we propose to perform a prostate MRI followed by a biopsy to evaluate for persistent/recurrent disease at 2 years after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage ≤ T2b according to the American Joint Commission on Cancer 6th Edition28
* PSA ≤ 15 ng/ml
* Gleason sum on biopsy ≤ 6 or 3+4=7
* Prostate volume ≤ 60 cc
* Willing to continue follow-up for at least two years

Exclusion Criteria:

* Prior hormone therapy
* Prior radiotherapy
* History of collagen vascular disease
* History of inflammatory bowel disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Chronic toxicity as assessed by the Common Toxicity Criteria Version 4.0 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Ennis, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- Saint Lukes-Roosevelt Hospital Center, New York, New York, United States